CLINICAL TRIAL: NCT00456950
Title: Detection of Vulnerable Plaque With Coronary Vessel Wall Magnetic Resonance Imaging
Brief Title: Magnetic Resonance Imaging of the Coronary Vessel Wall
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: T. Leiner, M.D., PhD, Dept. of Radiology, Maastricht University Hospital
Other Study IDs: MEC 04-272
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2009-09-24 (Estimated); Status verified 2009-09

CONDITIONS: Coronary Artery Disease
Keywords: coronary atherosclerosis; magnetic resonance imaging; vulnerable plaque
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Despite advances in prevention and treatment, clinical manifestations of atherosclerosis (e.g. myocardial infarction, stroke) remain the largest cause of mortality in the Western world. The occurrence of acute ischemic syndromes, including unstable angina and myocardial infarction, is highly associated with atherosclerotic plaque morphology.

Magnetic resonance (MR) imaging is able to noninvasively depict the lumen of coronary arteries without the need for ionizing radiation. In addition, MR imaging is able to generate soft-tissue contrast unlike any other imaging modality. It has been shown in the aorta and carotid artery that MR imaging is able to identify different atherosclerotic plaque components in vivo. Similar MR imaging techniques are becoming available to visualize the coronary arterial wall and preliminary studies have shown the feasibility of MR coronary vessel wall imaging in humans.

The overall aim of the current study is to identify in vivo MR coronary vessel wall and plaque features that are associated with acute coronary syndromes. This study is divided into 2 substudies:

1. Detection of atherosclerosis in the coronary vessel wall with contrast-enhanced MR imaging in patients with coronary artery disease and age-matched healthy volunteers.
2. Characterization of coronary vessel wall plaque morphology in patients with stable and unstable angina: validation of MRI with the current standard of reference intravascular ultrasound (IVUS).

ELIGIBILITY:
Inclusion Criteria:

* patients with (un)stable angina or non-ST-elevated myocardial infarction
* patients are scheduled for, or recently had X-ray coronary angiography
* healthy volunteers, no clinical history of coronary artery disease(control group for substudy 1)
* patients with non-ischemic heart disease, scheduled for X-ray coronary angiography (control group for substudy 2)
* informed consent

Exclusion Criteria:

* severe arrhythmia
* hemodynamic unstable patients
* contra-indications for MRI

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patients with (un)stable angina or non-st-elevated myocardial infarction: sample from dept. of cardiology
  * healthy volunteers: community sample
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2005-10; Primary Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Leiner, MD, PhD, Principal Investigator — Maastricht University Hospital
Locations (1):
- Maastricht University Hospital, Maastricht, Netherlands

REFERENCES:
- [Derived] Gerretsen SC, Kooi ME, Kessels AG, Schalla S, Katoh M, van der Geest RJ, Manning WJ, Waltenberger J, van Engelshoven JM, Botnar RM, Leiner T. Visualization of coronary wall atherosclerosis in asymptomatic subjects and patients with coronary artery disease using magnetic resonance imaging. PLoS One. 2010 Sep 29;5(9):e12998. doi: 10.1371/journal.pone.0012998. PMID 20927368